CLINICAL TRIAL: NCT00246935
Title: A Long-term Study of APTA-2217 in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Long-term Study of Safety and Efficacy of Roflumilast in Japanese Patients Older Than 40 Years With Chronic Obstructive Pulmonary Disease (APTA-2217-08)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APTA-2217-08
Record Dates: First submitted 2005-10-31; First posted 2005-11-01 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Phosphodiesterase 4 inhibitor; Roflumilast
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

INTERVENTIONS:
Drug: Roflumilast

SUMMARY:
The aim of this long-term study is to investigate the effect of roflumilast (APTA-2217) on the long-term safety in patients with chronic obstructive pulmonary disease (COPD) who completed the 24-week evaluation of study APTA-2217-06. Roflumilast will be administered orally once daily. The present study consists of a 28 weeks treatment period, and is an extension of the 24-week study APTA-2217-06 (registered study). The study will provide further long-term safety and efficacy data of roflumilast.

ELIGIBILITY:
Main inclusion criteria:

* Patients with chronic obstructive pulmonary disease (COPD)
* Written informed consent
* Patients who completed the 24-week evaluation of study APTA-2217-06

Main exclusion criteria:

* If patients required hospitalization or received emergency care for COPD exacerbation by the investigator (or sub-investigator) between the informed consent day and the starting day
* Patients with long-term oxygen therapy
* Serious diseases

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2005-05; Primary Completion 2007-01 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Long-term safety after 28 weeks treatment of Roflumilast (total 52 weeks, 24 weeks of study APTA-2217-06 followed by 28 weeks) .

SECONDARY OUTCOMES:
Efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (1):
- Nycomed in Japan and Mitsubishi Tanabe Pharma Corporation, Osaka, Japan

REFERENCES:
- See also: APTA-2217-08-RDS-2009-01-16.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4468&filename=APTA-2217-08-RDS-2009-01-16.pdf